CLINICAL TRIAL: NCT00212407
Title: New York Blood Center National Cord Blood Program
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Study NCT01656603 supersedes this study; FDA IND 6637
Sponsor: New York Blood Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 234
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2018-11-02 (Actual); Status verified 2018-10

CONDITIONS: Leukemia; Lymphoma; Genetic Disease; Severe Aplastic Anemia; Myelodysplasia
Keywords: Cord blood transplantation; bone marrow transplantation
MeSH Terms: conditions — Leukemia; Lymphoma; Genetic Diseases, Inborn; Anemia, Aplastic; Anemia, Refractory, with Excess of Blasts | interventions — Cord Blood Stem Cell Transplantation; Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Umbilical cord blood unit(s) transplant (Experimental): Transplantation of cryopreserved umbilical cord blood unit(s)
  Interventions: Biological: Umbilical Cord Blood Transplantation

INTERVENTIONS:
Biological: Umbilical Cord Blood Transplantation
  Other Names: One or more matched umbilical cord blood units for transplant

SUMMARY:
Umbilical cord blood is used as a source of hematopoietic stem cells for bone marrow reconstitution in patients who would be potential candidates for a bone marrow transplant from an unrelated marrow donor. The outcome of transplantation is obtained to assess cord blood myeloid and platelet engraftment, transplant related mortality, overall survival, graft vs. host disease and, for patients with leukemia, lymphoma or myelodysplasia, relapse.

DETAILED DESCRIPTION:
Umbilical cord blood donated to the New York Blood Center's National Cord Blood Program is collect, tested, processed, cryoprotected and frozen in liquid nitrogen for possible future transplantation to anyone who needs it. The Program has operated under a FDA IND exemption since 1996 and is licensed as a tissue bank by the New York State Department of Health.

Candidates for transplant are patients who disease requires bone marrow transplantation but who do not have a suitable related bone marrow donor. Most patients are those with high risk of refractory leukemia, lymphoma, myelodysplasia, severe aplastic anemia and certain genetic hematologic, immunologic and metabolic diseases.

Patients are treated at bone marrow transplant centers in the United States and in other countries with active marrow transplant programs. Because the NYBC Program operates under IND, patients must sign an informed consent for cord blood transplantation.

Transplant centers report on the transplant procedure (including immediate complications) and on transplant outcome at 3, 6 and 12 months post-transplant and annually thereafter. Data report to the New York Blood Center includes information about the patient's disease and pre-transplant conditioning regimen and post-transplant endpoints, primarily myeloid and platelet engraftment, transplant related mortality, overall survival, acute and chronic graft vs. host disease, relapse and other post-transplant complications such as infectious disease. The outcome data is used to assess safety and efficacy and will be used to apply for a license from the FDA.

ELIGIBILITY:
Inclusion Criteria:

* Candidates for bone marrow transplantation

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4476 (Actual)
Dates: Start 1993-02; Primary Completion 2011-11-10 (Actual); Study Completion 2011-11-10 (Actual)

PRIMARY OUTCOMES:
Engraftment | released prior to 12-1-2012
Treatment Related Mortality | released prior to 12-1-2012
Survival | released prior to 12-1-2012

SECONDARY OUTCOMES:
Graft vs. Host Disease | released prior to 12-1-2012
Relapse | released prior to 12-1-2012

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Rubinstein, M.D., Principal Investigator — New York Blood Center
Locations (1):
- New York Blood Center, New York, New York, United States

REFERENCES:
- See also: Click here for more information about the New York Blood Center National Cord Blood Program — http://www.nationalcordbloodprogram.org